CLINICAL TRIAL: NCT01078740
Title: Detection of Cystic Fibrosis Transmembrane Conductance Regulator CFTR) Activity in Rectal Tissues From Human Subjects
Brief Title: Detection of Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Activity in Rectal Tissues From Human Subjects
Status: Completed | Type: Observational
Sponsor: CF Therapeutics Development Network Coordinating Center (Network)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ICM001
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; cystic fibrosis transmembrane conductance regulator; biomarkers; Intestinal Current Measurement
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Rectal biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non-CF subjects: Rectal tissue obtained from study subjects without cystic fibrosis (CF) as part of scheduled colonoscopy/biopsies performed for clinical care
- CF subjects: Rectal tissue obtained from study subjects with cystic fibrosis (CF) in one of three ways:
  * Rectal biopsy as part of scheduled colonoscopy/biopsies performed for clinical care
  * Sigmoidoscopy/biopsy added onto a scheduled, unrelated procedure or surgery performed under general anesthesia
  * Sigmoidoscopy/biopsy performed for the sole purpose of obtaining rectal tissue for the current study

SUMMARY:
This is a pilot study. The purpose of the study is to facilitate the development of a new biomarker of cystic fibrosis transmembrane conductance regulator (CFTR) function using rectal tissue.

DETAILED DESCRIPTION:
CF research has advanced to the point where small molecule agents have been developed to overcome the underlying genetic defects caused by CFTR mutations.

There is a critical need to develop new sensitive biomarkers of CFTR function and biochemistry that can be used in early phase clinical trials to demonstrate biologic effects of investigative agents in vivo. Intestinal Current Measurement (ICM) from rectal biopsy samples is an assay that has been proven to be sensitive and specific for CFTR function. This method and site of investigation is particularly attractive, since CFTR is expressed at high levels in the rectum, it is not altered by disease manifestations, and the tissue can be studied ex vivo, providing more flexibility in the nature of the techniques to detect and quantify CFTR activity.

This study will aid in the development of new biomarkers in human rectal tissue for use in CF clinical trials. Testing compounds that are designed to restore function to disease-causing CFTR genes and proteins will provide an opportunity to improve and standardize techniques in the acquisition and measurement of CFTR activity in rectal biopsy specimens.

ELIGIBILITY:
1. Non-CF subjects

   Inclusion Criteria:
   * Male or female 18-75 years of age at enrollment
   * Undergoing colonoscopy for clinical care
   * Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

   Exclusion Criteria:
   * Any medical condition or laboratory values that in the opinion of the onsite principal investigator and/or collaborating gastroenterologist may place the subject at significant risk by undergoing the additional research related biopsies
   * Subjects with a history of radiation therapy to the rectum, prostate and/or pelvic area
2. CF subjects undergoing a surgical procedure for clinical care

   Inclusion Criteria:
   * Confirmed diagnosis of CF based on the following criteria: ∆F508 homozygous
   * Male or female 18 years of age or greater at enrollment
   * Patient undergoing planned colonoscopy or other surgical procedure and agrees to undergo sigmoidoscopy and biopsy
   * Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

   Exclusion Criteria:

   Any medical condition or laboratory values that in the opinion of the onsite principal investigator and/or collaborating gastroenterologist may place the subject at significant risk by undergoing the additional research related biopsies, including:
   * Significantly diseased distal rectal/gastrointestinal (GI) tissue (as judged by the collaborating gastroenterologist including radiation injury or history of radiation therapy to the rectum, prostate and/or pelvic area
   * Significant hemorrhoids or vascular abnormalities (as judged by the collaborating gastroenterologist)
   * Significant colonic infection (as judged by the collaborating gastroenterologist)
3. CF subjects undergoing sigmoidoscopy biopsy procedure for study purposes only

Inclusion Criteria:

* Confirmed diagnosis of CF based on the following criteria: ∆F508 homozygous
* Male or female 18 years of age or greater at enrollment
* Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study
* CBC, PT/PTT within acceptable range (see exclusion criteria for values) within 14 days of the procedure
* Negative pregnancy test (if applicable) completed within two (2) days of the procedure

Exclusion Criteria:

Any medical condition or laboratory values that in the opinion of the onsite principal investigator and/or collaborating gastroenterologist may place the subject at significant risk by undergoing the additional research related biopsies, including:

* Bleeding diathesis (platelets <50,000, INR >1.5)
* Anemia (hemoglobin <10 gm/dL, or hematocrit <30%
* White blood count >20,000
* Neutropenia (ANC <1,500) or lymphopenia (absolute lymphocyte count <1,500)
* Positive pregnancy test (if applicable)
* Breastfeeding
* Significantly diseased distal rectal/GI tissue that could place the study subject at risk by participating in the study (as judged by the collaborating gastroenterologist, such as significant hemorrhoids, vascular abnormalities, colonic infection, radiation injury or history of radiation therapy to the rectum, prostate and/or pelvic area)
* Use of drugs with significant risks of compromising immunity (oral steroid use > 20 mg/day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-CF subjects: Adults undergoing endoscopic procedures (colonoscopies) who meet the eligibility criteria.
  CF subjects: Adults with a diagnosis of CF who meet the eligibility criteria. CF subjects can include both patients who will be undergoing endoscopic (colonoscopies) and nonendoscopic procedures requiring anesthesia or sedation as a part of clinical care (e.g., sinus surgery, central line placement), or CF subjects not undergoing planned surgical/anesthetic procedures.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To develop and improve techniques to detect mature CFTR protein at the rectal cell membrane by performing rectal biopsies and ex-vivo Intestinal Current Measurement (ICM). | 24 hours

SECONDARY OUTCOMES:
To estimate the range of detectable CFTR activity among human rectal tissue of subjects with and without cystic fibrosis. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: JP Clancy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of North Carolina Hospitals, Chapel Hill, North Carolina